CLINICAL TRIAL: NCT06968949
Title: Collaborative Redesign of Implementation Strategies for the Brief Intervention for School Clinicians (BRISC)
Brief Title: Collaborative Redesign of Implementation Strategies for the Brief Intervention for School Clinicians
Acronym: BRISC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Eric Bruns, Professor, School of Medicine: Psychiatry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00019682; P50MH115837 (NIH)
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Anxiety Disorders; Depressive Symptoms; Mental Health Issue
Keywords: School Mental Health
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unadapted Brief Intervention for School Clinicians (BRISC; BR-O) (Active Comparator): Participants in this arm will receive unadapted Brief Intervention for School Clinicians (BRISC), a four-session engagement, brief intervention, and triage strategy targeting a range of mental health (e.g., anxiety, depression, past trauma) and other problems (academic, peer, family).
  Interventions: Behavioral: Unadapted Brief Intervention for School Clinicians (BRISC; BR-O)
- BRISC with Implementation Strategies Adapted for School Practitioners (BR-A) (Experimental): Participants in this arm will Brief Intervention for School Clinicians (BRISC) with implementation strategies adapted for school-employed practitioners (BR-A).
  Interventions: Behavioral: Brief Intervention for School Clinicians (BRISC) with Implementation Strategies Adapted for School-Employed Practitioners (BR-A)

INTERVENTIONS:
Behavioral: Unadapted Brief Intervention for School Clinicians (BRISC; BR-O) — BRISC is a four-session, individual engagement, assessment, brief intervention and triage strategy for youth age 13-18. BRISC provides a research-based approach to improving structure, efficiency, and effectiveness of school mental health via five elements: (1) Stepped care/tiered structure; (2) Culturally-informed engagement and motivation strategies;(3) Systematic problem-solving framework; (4) Modularized common elements approach; and (5) Structured assessment and monitoring.BRISC is hypothesized to operate on specific mechanisms that influence improvements in efficiency and clinical outcomes.
  Arms: Unadapted Brief Intervention for School Clinicians (BRISC; BR-O)
Behavioral: Brief Intervention for School Clinicians (BRISC) with Implementation Strategies Adapted for School-Employed Practitioners (BR-A) — BR-A is a version of the Brief Intervention for School Clinicians with implementation strategies (IS) adapted for delivery by in the education sector by school-employed practitioners. Although IS modifications will be determined by Study 1 activities, we anticipate that BR-A may include changes to training pacing or format (e.g., asynchronous e-learning modules and videos); adaptations to format/content of consultation; and/ or addition of other ISs to enhance skills development (e.g., development of a learning collaborative) and/or overcome organizational or system barriers (e.g., educational outreach, changes to regulations). Core components of BRISC will be retained in the BR-A condition.
  Arms: BRISC with Implementation Strategies Adapted for School Practitioners (BR-A)

SUMMARY:
Schools are the most common venue for youth mental health services, but school mental health (SMH) typically does not use evidence-based clinical interventions (CI), common elements of effective mental health, or effective implementation strategies. To address this gap, a multidisciplinary team developed the Brief Intervention for School Clinicians (BRISC), a four-session engagement, brief intervention, and triage strategy targeting a range of mental health (e.g., anxiety, depression, past trauma) and other problems (academic, peer, family). BRISC outperformed SMH usual care on engagement, treatment completion, and youth self-reported problem severity. Although there are many evidence-based SMH strategies such as BRISC, integration into practice is poor because accompanying implementation strategies are often absent, poorly defined, or insufficiently tailored to the education context.

DETAILED DESCRIPTION:
The investigators will evaluate the impact of original BRISC (BR-O) implementation versus adapted BRISC (BR-A) implementation for students referred to SMH on mental health outcomes (i.e., student top problems, anxiety, depression, mental health functioning). The investigators hypothesize:

H-1: In both BR-O and BR-A, more students will experience clinical improvement on mental health outcomes (i.e., top problems, anxiety, depression, mental health functioning) than deteriorate or remain unchanged.

H-2: BR-A will demonstrate noninferiority to BR-O on mental health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Clinician participants: Counselors will be included if they (a) provide school-based services; (b) have not previously received formal training in BRISC; and (c) are not actively receiving support to implement another intervention.
* Youth participants: Students must meet eligibility criteria for BRISC including (a) being in grades 9-12 and 13 years or older (b) receiving school mental health services

Exclusion Criteria:

* Anyone not meeting inclusion criteria.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Implementation Strategy Usability Scale (ISUS) | Post-training, End of Year 1
  Usability will be evaluated with the 10-item Implementation Strategy Usability Scale (ISUS), which is based closely on the well-validated System Usability Scale. Ratings are on a 1 to 5 scale and yield a total score from 0 to 100. Half the items are reverse scored; higher total scores reflect greater usability. The ISUS has good inter-item consistency (a = .83) and sensitivity. Research has also demonstrated that the original version of the ISUS (the SUS) functions similarly - and yields similar scores - for adults and youth.
Participant Responsiveness Scale (PRS) | Post-training, End of Year 1
  Engagement will be measured using the Participant Responsiveness Scale (PRS), an adapted version of the 12-item Patient Responsiveness Scale tailored to be developmentally appropriate for children aged 8 and above as well as adults. The PRS measures two factors, Participation and Enthusiasm. The original Patient Responsiveness Scale has demonstrated strong reliability (a = .86) and construct validity.
Intervention Appropriateness Measure (IAM) | Baseline, 3 months, 6 months
  The Intervention Appropriateness Measure (IAM) is a rigorously developed, pragmatic instrument with strong good internal consistency (a = .87) and test-retest reliability (a = .87).
Adoption | Baseline, 3 months, 6 months
  Adoption is operationalized as the initiation of a clinician first BR-0 or BR-A session at any point during study participation.
Reach | Baseline, 3 months, 6 months
  Reach will be calculated using adoption data as the percentage of clinicians caseloads receiving BR-O or BR-A.
Youth Top Problems (YTP) | Baseline, 3 months, 6 months
  The Youth Top Problems (YTP) assessment is an assessment in which youth and caregivers are asked to list the problems they were most concerned about. Upon completion of the list, respondents are asked to assign a severity rating for each problem by answering the questions: how big of a problem is this for you? (0 = not at all to 10 = very, very much). Respondents are then asked to identify which of the problems listed is the biggest problem right now? Which one is the most important to work on? Then the second and third most important until 3 top problems are identified. The YTP shows excellent concurrence with standardized assessments (Kappa ranging from .78 to .91), while also adding specificity for treatment targets (41% of caregivers-, and 79% of youth-identified top problems were not identified by an item amongst elevated standardized assessment subscales).
Therapeutic Alliance Scale for Adolescents (TASA) | Baseline, 3 months, 6 months
  Therapeutic Alliance Scale for Adolescents (TASA) is a widely used rating scale designed to measure the working alliance between clinicians and their adolescent clients. Youth and Counselor forms will be used. Both include 12 seven-point Likert Scale items covering three domains: bond, goals, and tasks.
Treatment Completion/Triage | End of study
  A measure of treatment efficiency, records will be reviewed of treatment disposition after 4 sessions, as well as triage to school/community services/supports.
Patient Health Questionnaire (PHQ-8 for Adolescent) | Baseline, 3 months, 6 months
  The Patient Health Questionnaire is one of the most used short depression measures. We will use the Adolescent adopted version of the PHQ-8, which removes the 9th item regarding suicide, which is commonly done in research settings where follow-up may be delayed; this has only minor effect on scoring and does not impact scoring interpretations. The PHQ features 8 items on a four-point scale (0=not at all, 1=several days, 2=more than half the days, 3=nearly everyday) with cutpoints for 5, 10, 15, and 20 representing mild, moderate, moderately severe, and severe levels of depressive symptoms. Four original validation studies were conducted on nearly 10,000 patients, and there have been multiple meta-analyses. Scores have been found valid, with sensitivity of 88% and specificity of 88% for a cutpoint of 10 has been found for Major Depressive Disorders.
Generalized Anxiety Disorder-7 scale (GAD-7) | Baseline, 3 months, 6 months
  Generalized Anxiety Disorder-7 scale (GAD-7) is a brief scale that queries about anxiety symptoms. Normative data for the GAD-7 included a large sample of adolescents aged 14-25 years (n = 634) that concluded the measure demonstrated age invariance, reliability, and internal consistency.
Columbia Impairment Scale (CIS) | Baseline, 3 months, 6 months
  The Columbia Impairment Scale (CIS) is a 13-item scale that measures adolescents level of adaptive functioning. The scale was used in the NIMH Methods for the Epidemiology of Child and Adolescent Mental Disorders (MECA) study and showed good reliability and validity. It is also correlated with other indicators of psychological distress and with standardized clinician ratings.
Quality of Life in Neurological Disorders Social Relations scale (Neuro-QOL) | Baseline, 3 months, 6 months
  The Quality of Life in Neurological Disorders Social Relations scale (Neuro-QOL) is a widely used 8-item measure of functioning in usual social roles, activities, and responsibilities. Factor analyses and Item Response Theory analyses have ensured broad information parameters without differential item functioning by demographics. Scale scores have been validated and normed on thousands of participants in the US general and clinical inpatient and outpatient settings, presenting with a variety of problem areas. Scores provide a T score with a mean of 50 and SD of 10, aligned with a variety of norming samples. An example item stem is : In the past 7 days I am able to do all of my regular family activities. Response options are on a scale of 1 to 5(1=never, 2=rarely, 3=sometimes, 4=often, 5=always).
Academic Progress Self-Report | Baseline, 3 months, 6 months
  Academic Progress Self-Report is a form successfully employed in other studies of school-based services by the research team to gauge academic success in areas such as homework completion, attendance, tardies, disciplinary action, and praise or discipline from school staff.

SECONDARY OUTCOMES:
BRISC External Rating Tool (BECT) | Baseline, 3 months, 6 months
  For each case, three recordings will be randomly selected from each BRISC treatment phase and coded for fidelity using the BRISC External Rating Tool (BECT).
Framework for Modifications and Adaptations of Evidence-Based Interventions | Baseline, 3 months, 6 months
  Recorded intervention sessions will be evaluated using the coding system for the Framework for Modifications and Adaptations of Evidence-Based Interventions (FRAME), the leading method for evaluating the nature of intervention adaptations

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bruns, Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: No